CLINICAL TRIAL: NCT01102192
Title: The Role of the Thymus in Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: Thymus in myasthenia gravis
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Myasthenia Gravis; Thymoma
Keywords: Myasthenia gravis; Thymoma; T-cells; Thymectomy
MeSH Terms: conditions — Myasthenia Gravis; Thymoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (serum, plasma), Thymoma tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Myasthenia gravis with thymoma: Myasthenia gravis with thymoma
- Myasthenia gravis without thymoma: Myasthenia gravis without thymoma
- Thymoma without Myasthenia gravis: Thymoma without Myasthenia gravis
- cardiac, or thyroid surgery: cardiac, or thyroid surgery

SUMMARY:
Although the association between thymic hyperplasia / thymoma and autoimmune myasthenia gravis has been known for some time, the question of causality remains uncertain. Recent research findings indicate, however, that especially in myasthenia patients with thymomas a non-physiological export of naive CD4 + T-cells can take place by the tumour and this could possibly play an important role in the pathogenesis of myasthenia gravis. The investigators want to analyse the functionality and specificity of t-cells generated in thymomas as well as the effect of thymectomy on the immune system.

DETAILED DESCRIPTION:
On one hand we want to perform a detailed analysis of the T-cells generated in thymomas in terms of their functional capacity and their specificity. We will analyse blood and thymoma tissue of patients with myasthenia gravis with thymona, patients with myasthenia gravis without thymona, and patients with thymona without myasthenia gravis.

Hypothesis: The T-cells which are generated in the thymoma in thymoma-associated myasthenia gravis can be differentiated from T-cells which are generated in normal thymoma tissue with regard to functionality and T-cell receptor specificity. This non-physiological T-cell maturation might be the cause for the formation of auto-antibodies.

On the other hand we want to examine the effects of thymectomy on the immune system in the context of myasthenia gravis. We will analyse blood and thymoma tissue of patients with myasthenia gravis with thymona, patients with myasthenia gravis without thymona, patients with thymona without myasthenia gravis and patients with cardiac, or thyroid surgery.

Hypothesis:

1. Thymectomy in patients with myasthenia gravis leads to a reduced number of auto-reactive, e.g. Acetylcholine receptor (ACh-R)-specific T cells. In contrast, T-cells with other specifities, for example against CMV or tetanus, are not affected.
2. The non-physiological export of thymocytes from thymomas leads to a significant shift in leukocyte populations in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with compelling indications for thymectomy due to thymoma (with or without myasthenia gravis), Or
* Patients with elective indication for thymectomy due to thymoma without myasthenia gravis
* Patients with indication for a heart or thyroid surgery, in which for op-technical reasons, a (partial) resection of the thymus is performed.
* Signed informed consent form
* Age > 17 Years

Exclusion Criteria:

* Other immunological diseases such as rheumatoid arthritis, multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without Mystenia gravis (with and without thymona) and patients with an indication for a heart or thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite University (Dept of Neurology & NeuroCure Clinical Research Center NCRC), Berlin, Germany

REFERENCES:
- [Result] Kohler S, Keil T, Alexander T, Thiel A, Swierzy M, Ismail M, Ruckert JC, Meisel A. Altered naive CD4+ T cell homeostasis in myasthenia gravis and thymoma patients. J Neuroimmunol. 2019 Feb 15;327:10-14. doi: 10.1016/j.jneuroim.2019.01.005. Epub 2019 Jan 11. PMID 30686546
- [Result] Kohler S, Keil TOP, Hoffmann S, Swierzy M, Ismail M, Ruckert JC, Alexander T, Meisel A. CD4+ FoxP3+ T regulatory cell subsets in myasthenia gravis patients. Clin Immunol. 2017 Jun;179:40-46. doi: 10.1016/j.clim.2017.03.003. Epub 2017 Mar 9. PMID 28286113
- [Result] Kohler S, Keil TO, Swierzy M, Hoffmann S, Schaffert H, Ismail M, Ruckert JC, Alexander T, Hiepe F, Gross C, Thiel A, Meisel A. Disturbed B cell subpopulations and increased plasma cells in myasthenia gravis patients. J Neuroimmunol. 2013 Nov 15;264(1-2):114-9. doi: 10.1016/j.jneuroim.2013.09.006. Epub 2013 Sep 18. PMID 24099983